CLINICAL TRIAL: NCT06846008
Title: The Effectiveness of a Coach-Focused Intervention on Preventing Acute Severe Knee Injuries in Amateur Football Players: A Cluster Randomized Superiority Trial
Brief Title: The Effectiveness of a Coach-Focused Intervention on Preventing Knee Injuries in Amateur Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APPI2-MSK-2025-KNIPS_2.0
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Knee Injuries
Keywords: knee injury; injury prevention training; football; coaches; players
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injury prevention training (Experimental): Evidence-based injury prevention training programs and exercises will be send weekly to participants in the intervention arm.
  Additionally, participants in the intervention arm will be encouraged to access a study specific online platform containing information, inspiration, pep-talks and posters on injury prevention training.
- Usual practice (Active Comparator): Usual training
  Interventions: Other: Usual Practice

INTERVENTIONS:
Behavioral: Ahead of the Game — Evidence-based injury prevention training programs and exercises will be send weekly to participants in the intervention arm.
  Additionally, participants in the intervention arm will be encouraged to access a study specific online platform containing information, inspiration, pep-talks and posters on injury prevention training.
Other: Usual Practice — Usual training
  Arms: Usual practice

SUMMARY:
The goal of this clinical trial is to find out if a coach-focused intervention can help prevent sudden-onset, severe knee injuries in youth and senior amateur football players. The main question it aims to answer is:

Does a coach-focused intervention reduce the number of sudden-onset, severe knee injuries? Researchers will compare a coach-focused intervention, designed to help coaches to use effective injury prevention training, to usual football practice to see if the intervention can prevent sudden-onset, severe knee injuries in football players.

Participants will:

Either receive weekly information and motivation on effective injury prevention training or continue their usual football practice for 14 weeks.

All will receive a weekly text message with a survey link to report any sudden-onset knee injuries among their players for 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Coach or manager at Danish amateur football teams at levels from under 14 (U14) years to senior teams.
2. Minimum 18 years of age.
3. Access to a mobile phone and computer.

Exclusion Criteria:

1. Limited Danish language skills, which prevents full understanding of the provided material and questionnaires.
2. Affiliation to teams playing under a license ranking by the Danish Football Association where training by a physical trainer is required according to the license criteria of the Danish Football Association).
3. Affiliation solely with old boys'/girls' teams (where the players have to be aged 32 and 29 , respectively, in the current season ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of acute severe knee injuries in players. | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in incidence of acute severe knee injuries (>28 time-loss days from training and matches) per 1000 hours of player exposure in players belonging to coaches in the intervention group compared with players belonging to coaches in the control group (usual practice) throughout the intervention period.

SECONDARY OUTCOMES:
Incidence of acute knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in incidence of all acute knee injuries (from minimal (1-3 days lost) to severe (>28 time-loss days from training or match)) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Incidence of acute minimal knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in incidence of acute minimal knee injuries (1-3 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Incidence of acute mild knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in incidence of acute mild knee injuries (4-7 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Incidence of acute moderate knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in incidence of acute moderate knee injuries (8-28 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Time-loss days of acute knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in burden of all acute knee injuries (the total number of time loss days from minimal (1-3 time-loss days) to severe (>28 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Time-loss days of acute minimal knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in burden of acute minimal knee injuries (1-3 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Time-loss days of acute mild knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in burden of acute mild knee injuries (4-7 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Time-loss days of acute moderate knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in burden of acute moderate knee injuries (8-28 time-loss days from training or match) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.
Time-loss days of acute severe knee injuries | From baseline to end of the intervention, 14 weeks after baseline.
  The difference in burden of acute and severe knee injuries (> 28 time-loss days from training or matches) per 1000 hours of player exposure in players belonging to coaches in the intervention group versus players belonging to coaches in the control group (usual practice) throughout the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bandak, PhD, Study Chair — The Parker Institute
Locations (1):
- The Parker Institute, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD can upon rasonable request to the investigator be shared.